CLINICAL TRIAL: NCT00480532
Title: A Study of Continuous Oral Contraceptives and Doxycycline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeffrey Jensen, MD MPH, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHSU FAMPLAN 2907
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Contraceptives, Oral
Keywords: birth control; continuous contraception; break-through bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — lybrel; Ethinyl Estradiol; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Doxycycline 100bid x5 days (Experimental)
  Interventions: Drug: Lybrel; Drug: Doxycycline; Drug: Doxycycline 100bid x5 days at the time of bleeding
- placebo bid x 5 days (Placebo Comparator)
  Interventions: Drug: Lybrel; Drug: Placebo
- Subantimicrobial doxycycline daily (Experimental)
  Interventions: Drug: Oracea; Drug: Subantimicrobial doxycycline daily
- placebo daily (Placebo Comparator)
  Interventions: Drug: placebo daily

INTERVENTIONS:
Drug: Lybrel — All women enrolled in the study will take the same daily low dose oral contraceptive (20-mcg EE/90 mcg LNG) dosed in a continuous fashion.
  Other Names: Lybrel (20-mcg Ethinyl Estradiol (EE)/90 mcg Levonorgestrel (LNG)
  Arms: Doxycycline 100bid x5 days; placebo bid x 5 days
Drug: Doxycycline — 100 mg orally twice a day for five days starting on the first day of breakthrough bleeding. This regimen will be repeated if bleeding persists or recurs seven days after completing five-day course of doxycycline.
  Arms: Doxycycline 100bid x5 days
Drug: Oracea — 40-mg tablet daily for 84 days
  Arms: Subantimicrobial doxycycline daily
Drug: Placebo — Placebo pill orally twice a day for five days starting on the first day of breakthrough bleeding. This regimen will be repeated if bleeding persists or recurs seven days after completing five-day course of placebo
  Arms: placebo bid x 5 days
Drug: Doxycycline 100bid x5 days at the time of bleeding — Doxycycline 100 mg orally twice a day for five days starting on the first day of breakthrough bleeding. This regimen will be repeated if bleeding persists or recurs seven days after completing five-day course of doxycycline
  Arms: Doxycycline 100bid x5 days
Drug: Subantimicrobial doxycycline daily — Subantimicrobial dose doxycycline 40mg daily for the first 84 days of the study
  Arms: Subantimicrobial doxycycline daily
Drug: placebo daily — Placebo daily for the first 84 days of the study
  Arms: placebo daily

SUMMARY:
The purpose of this study is to learn if the study drug, doxycycline, can decrease the amount of unplanned vaginal bleeding that women commonly experience when taking combined oral contraception (COC)- pills with estrogen and progestin - in a continuous fashion - no hormone-free week. The study drug, doxycycline, is an antibiotic used commonly for many conditions (i.e. acne, Chlamydia infections, pneumonia) and can be safely used on a daily basis. Doxycycline has been shown to decrease unplanned vaginal bleeding in progestin-only contraception but has not been studied in combined hormonal contraception.

DETAILED DESCRIPTION:
We intend to conduct a prospective, randomized, placebo controlled, double blind study at Oregon Health and Science University. This study will be conducted over four 28-day cycles (112 days of active COC hormone). All women enrolled in the study will take the same daily low dose COC. This protocol will be divided into two studies, a bleeding study and an endometrial biopsy study, each with two treatment arms; typical dose doxycycline (Arm 1), and controlled release subantimicrobial dose doxycycline (CRSD)(Arm 2).

The first arm (Arm 1) of this study will constitute the typical dose doxycycline arm. In this arm, there will be two study groups. Group 1, the treatment group, will take doxycycline 100 mg orally twice a day for five days starting on the first day of bleeding if breakthrough bleeding occurs. The control group will take a placebo orally twice a day for five days starting on the first day of bleeding if breakthrough bleeding occurs. After three months, both groups will stop doxycycline (or placebo) and will continue on a COC alone for the remaining 28 days of the study.

The second arm (Arm 2) of the study will constitute the controlled release subantimicrobial dose doxycycline (CRSD doxycycline)arm. Subjects in this arm of the study will be divided into Group 3 and Group 4. Group 3 will take CRSD doxycycline (40mg) daily for three months. Group 4 will take a daily placebo. Similarly to the first arm of the trial, after three months, both groups will stop doxycycline (or placebo) and will continue in a COC alone for the remaining 28 days of the study.

This study also includes a endometrial biopsy sub-study: At the time of recruitment we will identify participants who are willing to undergo endometrial biopsy during the study period. These subjects will constitute a separate cohort who will enroll in the prospective, randomized, double blind, placebo controlled endometrial biopsy study.

ELIGIBILITY:
Inclusion Criteria:

* General good health
* Willing and able to agree to randomization and sign informed consent
* Currently having regular menstrual cycles (24-36 days), with combined cyclic hormonal method (COCs, Nuva Ring, Ortho Evra), without intermenstrual bleeding in last 2 years.

Exclusion Criteria:

* Intrauterine device (IUD) in place
* Abnormal pap smear that has not been treated or followed up
* Those with hypersensitivity reactions to doxycycline or any of the tetracyclines
* Use of depomedroxyprogesterone acetate within 9 months of the start of the study.
* Use of hormonal medications (excluding cyclic contraceptives and plan B) within 2 months of the start of the study.
* Any one unwilling to keep a daily menstrual diary or otherwise unwilling to follow the study criteria
* Currently taking medications that interfere with COCs (rifampin, carbamazepine, St. Johns wort)
* Currently has a progestin implant
* Positive Gonorrhea or Chlamydia cultures at enrollment examination
* Smoking more than 5 cigarettes per month
* Any medical condition that is a contraindication to the use of COCs in accordance with product labeling including:

  * History of thrombophlebitis, deep venous thrombosis, thrombogenic vasculopathies, thrombogenic rhythm disorders or thromboembolic disorders
  * Current or past history of cerebrovascular or coronary artery disease
  * Scheduled major surgery in the next six months with prolonged immobilization
  * Diabetes with vascular involvement
  * Headache with focal neurologic symptoms
  * Uncontrolled hypertension
  * Suspected or known carcinoma of the breast or personal history of breast cancer
  * Carcinoma of the endometrium or other known or suspected estrogen dependent neoplasms
  * Undiagnosed genital bleeding
  * History of cholestatic jaundice of pregnancy or cholestatic jaundice with prior oral contraceptive use
  * Hepatic adenoma or carcinoma or active liver disease if liver function has not returned to normal
  * Known or suspected pregnancy
  * Hypersensitivity to estrogen or progesterone containing products

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2007-05; Primary Completion 2010-01 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T Jensen, M.D, MPH, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - University of Hawaii (UH), Honolulu, Hawaii
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Result] Kaneshiro B, Edelman A, Carlson N, Morgan K, Nichols M, Jensen J. Treatment of unscheduled bleeding in continuous oral contraceptive users with doxycycline: a randomized controlled trial. Obstet Gynecol. 2010 Jun;115(6):1141-1149. doi: 10.1097/AOG.0b013e3181e0119c. PMID 20502283
- [Result] Kaneshiro B, Edelman A, Carlson NE, Nichols M, Forbes MM, Jensen J. A randomized controlled trial of subantimicrobial-dose doxycycline to prevent unscheduled bleeding with continuous oral contraceptive pill use. Contraception. 2012 Apr;85(4):351-8. doi: 10.1016/j.contraception.2011.08.006. Epub 2011 Sep 28. PMID 22067758
- See also: Women's Health Research Unit website — http://www.ohsuwomenshealth.com/research/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at Oregon Health and Science University (OHSU) and University of Hawaii (UH
Groups:
- Placebo (Treatment): Placebo (for treatment portion of the study)
- Doxy (7 Day Treatment Arm): Doxycycline 100 mg po bid x 7 days taken when bleeding occurred
- Placebo (Prevention): Placebo for prevention portion of the study
- Subantibmicrobial Dose Doxy: Doxycycline 40mg (sustained release) once daily for 84 days
Period: Overall Study
Arm/Group | Placebo (Treatment) | Doxy (7 Day Treatment Arm) | Placebo (Prevention) | Subantibmicrobial Dose Doxy
Started | 33 | 33 | 33 | 32
Completed | 31 | 29 | 29 | 31
Not Completed | 2 | 4 | 4 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 3 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Treatment) | Doxy (7 Day Treatment Arm) | Placebo (Prevention) | Subantibmicrobial Dose Doxy | Total
Number analyzed (Participants) | 33 | 33 | 33 | 32 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 1
  Between 18 and 65 years | 33 | 33 | 33 | 31 | 130
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (6.6) | 27.5 (6.8) | 27.8 (5.4) | 28.6 (6.1) | 28.0 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 33 | 32 | 131
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 33 | 32 | 131

OUTCOME MEASURES:

1. Primary Outcome: Differences in Bleeding Patterns Between Study Groups.
Description: number of days of bleeding and spotting, self reported on calendar
Time Frame: The outcome was also assessed for day 1 to 84
Population: All participants analyzed in the groups to which they were randomized except for 1 subject in prevention placebo group who was erroneously enrolled although she did not meet enrollment entry criteria
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo (Treatment) | Doxy (7 Day Treatment Arm) | Placebo (Prevention) | Subantibmicrobial Dose Doxy
Number analyzed (Participants) | 33 | 33 | 32 | 32
days | 26.72 (4.89) | 31.86 (5.08) | 25.69 (3.24) | 18.84 (3.30)

2. Secondary Outcome: Subject Satisfaction.
Description: measured using 100 mm visual analog scale. anchors of "not at all satisfied" (0mm) "extremely satisfied" (100mm)
Time Frame: Assessed on day 112 of the study (the end of the study period). This outcome does not represent a change from baseline. It was assessed at the end of the study period.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo (Treatment) | Doxy (7 Day Treatment Arm) | Placebo (Prevention) | Subantibmicrobial Dose Doxy
Number analyzed (Participants) | 33 | 33 | 32 | 32
mm | 63.9 (41.1) | 64.2 (33.0) | 72.0 (30.9) | 67.0 (35.3)

3. Secondary Outcome: Subject Compliance
Description: measured by self report of pill intake on daily diary (yes/no), and reported as percentage with no missed pills over entire study
Time Frame: Assessed on day 112 of the study (the end of the study period). The outcome reflects the number of subjects who did not miss pills during the entire 112 day study. It does not represent a change from baseline.
Measure: Number; unit: number of participants with no missed pi
Arm/Group | Placebo (Treatment) | Doxy (7 Day Treatment Arm) | Placebo (Prevention) | Subantibmicrobial Dose Doxy
Number analyzed (Participants) | 33 | 33 | 32 | 32
number of participants with no missed pi | 25 | 21 | 19 | 20

ADVERSE EVENTS:
Arm/Group | Placebo (Treatment) | Doxy (7 Day Treatment Arm) | Placebo (Prevention) | Subantibmicrobial Dose Doxy
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/32 | 0/32

LIMITATIONS AND CAVEATS:
Treatment Arm: Subjects had difficulty understanding when to start and stop treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No